CLINICAL TRIAL: NCT00391664
Title: Gynecologic Cancer Survivorship Survey
Brief Title: Questionnaire Study for Gynecological Cancer Survivors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: Walter Reed Army Medical Center (U.S. Federal Agency); Ohio State University (Other)
Organization: Walter Reed Army Medical Center (U.S. Federal Agency)
Other Study IDs: 05-44025
Record Dates: First submitted 2006-10-23; First posted 2006-10-24 (Estimated); Last update posted 2008-06-30 (Estimated); Status verified 2008-06

CONDITIONS: Endometrial Neoplasms; Ovarian Neoplasms; Uterine Cervical Neoplasms; Vulvar Neoplasms; Vaginal Neoplasms; Genital Neoplasms, Female
Keywords: Endometrial cancer; Ovarian Cancer; Cervical Cancer; Genital Cancer; Vulvar Cancer; Vaginal Cancer; Other Gynecological Cancers
MeSH Terms: conditions — Endometrial Neoplasms; Ovarian Neoplasms; Uterine Cervical Neoplasms; Vulvar Neoplasms; Vaginal Neoplasms; Genital Neoplasms, Female

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Behavioral: Psychosocial

SUMMARY:
The purpose of this study is to evaluate the quality of life of long-term gynecologic cancer survivors.

DETAILED DESCRIPTION:
Since the early 1970s, death rates for the major gynecological tumors have significantly declined, with a reduction of 42% for endometrial, 49% for cervix, 27% for vagina and vulva, and 11% for ovarian cancer. Thus, of the approximately 82,000 new gynecologic cases each year, more women will be living and, necessarily be forced to cope with psychological or behavioral morbidity. Psychosocial data on cancer patients portray significant fear and anxiety with diagnosis and treatments and the potential for high levels of psychological and sexual morbidity. While many studies have been done investigating sexual outcomes, little data is available on basic domains of quality of life, i.e. emotional or social adjustment, occupational outcomes, or aspects of physical health that might influence quality of life for gynecologic cancer survivors. There is a need for basic descriptive research in these areas, particularly in investigations that include representative samples from differing socioeconomic and racial/ethnic groups.

The goal of the proposed study is to evaluate quality of life in long-term gynecologic cancer survivors. The specific aims are to:

1. Describe quality of life (both mental health and physical functioning components), stress, and sexual functioning among survivors of gynecologic malignancies and
2. Describe differences between disease site groups (i.e. cervical, endometrial, ovarian, and vulva).

It has been shown with other cancer groups that improvements in mood and coping can be achieved with brief, cost effective interventions (e.g. ten therapy hours with delivery in a group format). These are multi-modal interventions with stress reduction, disease/treatment information, cognitive behavioral coping strategies, and social support. There is suggestive evidence that disease specific interventions, such as including sexual therapies for gynecologic patients, can result in improvements as well. Research focus on these issues is aided by the availability of reliable and valid strategies to assess both quality of life (SF-36; FACT) and sexuality. Before clinical trials are undertaken, research must provide a comprehensive assessment of quality of life for gynecologic cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Female participants diagnosed with gynecologic cancer
* Participants between the ages of 20 and 75 years old, inclusive
* Participants previously treated for all stages (I-IV) of the following cancers: cervix; endometrium; ovary; vulva; vagina; and other genital cancers
* Participants receiving treatment for their primary cancer in the past 2-10 years

Exclusion Criteria:

* Male participants
* Participants with major psychoses (e.g. organic brain syndrome; schizophrenia; bipolar disorder; or mental retardation).
* Participants with significant hearing deficit
* Participants with prior non-gynecologic cancer diagnosis
* Participants who refused all forms of cancer treatment, whether standard of care or experimental.
* Participants with deficient ability to read/speak English
* Participants residing >90 miles from the research site
* Participants diagnosed with dementia
* Participants diagnosed with pregnancy

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2006-02; Study Completion 2011-02

CONTACTS AND LOCATIONS:
Overall Officials: Barbara L Andersen, PhD, Study Director — Ohio State University; LTC G. Larry Maxwell, MD, Principal Investigator — Walter Reed Army Medical Center
Locations (2):
- United States (2):
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Ohio State University, Columbus, Ohio